CLINICAL TRIAL: NCT04229186
Title: Pilot Study About Extra Virgin Oil "Coratina" (Evoo-c) in Mild Cognitive Impairment (MCI) and Alzheimer's Disease (AD) Patients (EVOO-c in MCI/AD)
Brief Title: Pilot Study About Extra Virgin Olive Oil "Coratina" in Mild Cognitive Impairment and Alzheimer's Disease Patients
Acronym: EVOCAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bari Aldo Moro (Other)
Collaborators: Med & Food and Schena Foundation (Unknown)
Responsible Party: Principal Investigator, Maria Trojano, Full Professor, University of Bari Aldo Moro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 5752
Record Dates: First submitted 2019-09-23; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Neurodegenerative Diseases
Keywords: Mild Cognitive Impairment; Alzheimer's Disease; Extra Virgin Olive Oil
MeSH Terms: conditions — Neurodegenerative Diseases; Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with assumption of EVOO-C (Experimental): 12 patients with Mild Cognitive Impairment or Mild Alzheimer's Disease will receive 10 mg EVOO-C
  Interventions: Dietary Supplement: EVOO-C
- Patients with assumption of ROO (Experimental): 12 patients with Mild Cognitive Impairment or Mild Alzheimer's Disease will receive 10 mg ROO
  Interventions: Dietary Supplement: ROO

INTERVENTIONS:
Dietary Supplement: EVOO-C — Each patient will consume 10 mg total daily amount EVOO-C
  Arms: Patients with assumption of EVOO-C
Dietary Supplement: ROO — Each patient will consume 10 mg total daily amount ROO
  Arms: Patients with assumption of ROO

SUMMARY:
Alzheimer's Disease is a neurodegenerative disease age related caused by neurofibrillary tangles misfolding and Beta-amyloid protein accumulation. In the last decade several findings showed the role of biophenols present in diary intake such as extra virgin olive oil as potential antagonist of neurodegeneration. Two population studies (The Seven Countries Study and Three-City-Study) and four clinical trials (PREDIMED, PREDIMED - NAVARRA, ACTRIN and ISRCTN) have already suggested that mediterranean diet or other diets supplemented with extra virgin olive oil could improve cerebral performance.

DETAILED DESCRIPTION:
24 MCI or Alzheimer's Disease patients will be recruited and randomised; 12 of them will receive extra virgin olive oil "coratina" (EVOO-C); 12 of them will receive biophenol low dose olive oil (ROO). Each patient will consume a total amount of 10 mg olive oil in a year (12 months). Clinical assessement will be based on:

* neurological examination (T0, T6, T12);
* cardiological examination (T0, T12): a supra-aortic vessels and brachial artery ecocolordoppler will be performed;
* ophthalmological evaluation (T0, T12): a optic coherence tomography will be performed;
* neuropsychological assessment (T0, T12);
* nutritional assessement(T0, T3, T6, T9, T12).

Each subject will perform:

* brain MRI (T0, T12);
* Beta Amyloid Positron Emission Tomography (T0, T12) A lumbar puncture will be ruled as well (T0) and markers of neurodegeneration (Beta-amyloid 1 - 42, total tau protein, fosfo-tau, Brain Derived Neurotrophic Factor (BDNF), Neurofilament (NFL) will be quantified); Renal, hepatic and nutritional status will be assessed 3 times in 12 months (T0, T6, T12).

ELIGIBILITY:
Inclusion Criteria:

* MCI diagnosis in the last month prior the recruitment;
* Clinical Dementia Rating Scale - Global Score (CDR - GS) 0,5 and Mini Mental Examination 24 - 27;

Exclusion Criteria:

* smoke;
* hypertension;
* diabetes;
* positive history of stroke, epilepsy or cardiac disease;
* BMI > 30;
* depression or other psychiatric disturbances;
* low compliance to medical interventions;
* positive history of olive oil allergy or intolerance;
* positive history of chronic inflammatory intestinal disease or malabsorption;
* positive history of maculopathy or retinopathy;
* MRI leukoaraiosis II-III grade Fazekas or MRI lacunar infarctions

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the change of cerebral performance after olive oil supplementation. | Change from baseline MMSE score at 12 months
  The change of cerebral performance will be documented by neuropsychological assessement with Minimental State Examination (MMSE) (total score)
Evaluate the change of nutritional parameters after olive oil supplementation | Change from baseline BMI at 3 months, from baseline BMI at 6 months, from baseline BMI at 12 months
  Weight and height will be combined to report BMI in Kg/m^2. Nutritional assessment will be measured comparing the variation of BMI of each patient during the follow up.
Evaluate the change of neurodegenerative biomarkers after olive oil supplementation. | Change from baseline neurodegenerative biomarkers at 3 months, from baseline neurodegenerative biomarkerse at 6 months, from baseline neurodegenerative biomarkers at 12 months
  Neurodegenerative biomarkers will be tested with blood samples and with cerebrospinal fluid analisys (cerebrospinal level of Beta-amiloid, Tau and phospotau, BDNF (pg/mL; blood level of BDNF e NFL (pg/mL))
Evaluate the change of neurodegenerative biomarkers after olive oil supplementation. | Change from baseline neurodegenerative biomarkers at 12 months
  Neurodegenerative biomarkers will be tested with blood samples and with cerebrospinal fluid analysis (cerebrospinal level of Beta-amyloid, Tau and phosphotau, BDNF (pg/mL; blood level of BDNF e NFL (pg/mL))
Evaluate the change of optic nerve and macula thickness after olive oil supplementation. | Change from baseline optic nerve and macula thickness at 12 months
  Ocular computerized tomography will be performed and layer of retinal nerve fiber will be measured (micron)
Evaluate the change of cortical thickness with brain MRI after olive oil supplementation. | Change from baseline at 12 months
  Brain MRI will be performed to assess cortical thickness using Normalized Thickness Index (NTI)
Evaluate the change of brain amyloid plaque load (BAPL) after olive oil supplementation. | Change from baseline BAPL at 12 months
  Beta amyloid positron emission tomography will be performed measuring a index called BAPL.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao LN, Long HW, Mu Y, Chew LY. The toxicity of amyloid beta oligomers. Int J Mol Sci. 2012;13(6):7303-7327. doi: 10.3390/ijms13067303. Epub 2012 Jun 13. PMID 22837695
- [Background] Coppola G, Di Renzo A, Ziccardi L, Martelli F, Fadda A, Manni G, Barboni P, Pierelli F, Sadun AA, Parisi V. Optical Coherence Tomography in Alzheimer's Disease: A Meta-Analysis. PLoS One. 2015 Aug 7;10(8):e0134750. doi: 10.1371/journal.pone.0134750. eCollection 2015. PMID 26252902
- [Background] Fazekas F, Chawluk JB, Alavi A, Hurtig HI, Zimmerman RA. MR signal abnormalities at 1.5 T in Alzheimer's dementia and normal aging. AJR Am J Roentgenol. 1987 Aug;149(2):351-6. doi: 10.2214/ajr.149.2.351. PMID 3496763
- [Background] Jack CR Jr, Holtzman DM. Biomarker modeling of Alzheimer's disease. Neuron. 2013 Dec 18;80(6):1347-58. doi: 10.1016/j.neuron.2013.12.003. PMID 24360540
- [Background] Caminiti SP, Ballarini T, Sala A, Cerami C, Presotto L, Santangelo R, Fallanca F, Vanoli EG, Gianolli L, Iannaccone S, Magnani G, Perani D; BIOMARKAPD Project. FDG-PET and CSF biomarker accuracy in prediction of conversion to different dementias in a large multicentre MCI cohort. Neuroimage Clin. 2018 Jan 28;18:167-177. doi: 10.1016/j.nicl.2018.01.019. eCollection 2018. PMID 29387532